CLINICAL TRIAL: NCT07386405
Title: Italian Version of KOOS-ACL (Knee Injury and Osteoarthritis Outcomes Score - Anterior Cruciate Ligament): Translation, Cross-cultural Adaptation and Validation
Brief Title: Validation and Cultural Adaptation of the KOOS-ACL Scale for the Italian Population
Acronym: VACKP
Status: Not yet recruiting | Type: Observational
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Other Study IDs: KOOS-ACL Validation (VACKP)
Record Dates: First submitted 2026-01-27; First posted 2026-02-04 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Scale Reliability Validity; ACL Injury; Validation and Cultural Adaptation of a Scale; PROMs
Keywords: scale reliability; ACL; KOOS-ACL; PROMs
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PROMS submition — KOOS ACL submission to validate and transalte the scale for italian people

SUMMARY:
Submission of the KOOS ACL questionnaires in Italian for the purpose of validation and cultural adaptation of the KOOS-ACL scale for the Italian population.

ELIGIBILITY:
Inclusion Criteria:

* Patient age 18 years or older
* Patients who are native Italian speakers
* Patients undergoing anterior cruciate ligament reconstruction of the knee
* Patients who have understood and signed the informed consent to participate in the study.
* Patients who are able to understand the study conditions and participate for the entire duration

Exclusion Criteria:

* Patients unable to understand the text in Italian
* Patients undergoing knee replacement surgery, corrective osteotomies, or osteosynthesis of knee fractures.
* Patients who are drug addicts, alcoholics, suffer from psychiatric disorders, or have any clinical conditions that could compromise the success of the questionnaire.
* Patients with orthopedic conditions of other origins

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of anterior cruciate ligament injury, undergoing or being considered for ACL reconstruction surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
validated translation and cultural adaptation of the KOOS-ACL scale in Italian. | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Clinico San Siro, Milan, Italy

IPD SHARING:
Plan to Share IPD: No